CLINICAL TRIAL: NCT02895659
Title: Fluid Management in Patients Undergoing Cardiac Surgery - Effects of an Acetate Versus Lactate Buffered Balanced Infusion Solution on Hemodynamic Stability, a Randomized Controlled Double-blind Trial
Brief Title: Fluid Management in Patients Undergoing Cardiac Surgery
Acronym: Hemacetat
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20160804.1.3
Record Dates: First submitted 2016-08-30; First posted 2016-09-12 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Critical Illness
Keywords: fluid management; critical illness; hemodynamics; buffered infusates
MeSH Terms: conditions — Critical Illness | interventions — Norepinephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ringer lactate (Active Comparator): Fluid resuscitation will be performed with lactated Ringers during the perioperative period. Perioperative hemodynamic management will be performed according to a specified treatment protocol.
  Interventions: Procedure: perioperative hemodynamic management with vasoactive medications (norepinephrine, adrenaline ect)
- Ringer acetate (Active Comparator): Fluid resuscitation will be performed with acetated Ringers during the perioperative period. Perioperative hemodynamic management will be performed according to a specified treatment protocol.
  Interventions: Procedure: perioperative hemodynamic management with vasoactive medications (norepinephrine, adrenaline ect)

INTERVENTIONS:
Procedure: perioperative hemodynamic management with vasoactive medications (norepinephrine, adrenaline ect) — Perioperative hemodynamic management will be performed according to a specified treatment protocol.

SUMMARY:
Background: Currently used crystalloid solutes have a variable composition and may therefore influence acid-base status, intra- and extracellular water content and plasma electrolyte compositions and have a major impact on organ function and outcome. Despite continuing evaluation no superiority of one particular type of fluid has been reached so far. To the best of the investigators' knowledge no study in humans has ever assessed whether the type of crystalloid fluid given for fluid resuscitation in patients undergoing cardiac surgery has an impact on hemodynamic stability and cardiac function so far. Nonetheless in the animal model it was shown that the choice of crystalloid fluid may greatly influence cardiac performance

Primary Aim: In this study the investigators want to clarify whether a balanced type acetate-buffered fluid solution in patients undergoing cardiac surgery is associated with better hemodynamic stability and cardiac function than a lactate-buffered crystalloid solute.

ELIGIBILITY:
Inclusion Criteria:

* Elective single heart valve replacement
* Elective double valve replacement
* Elective single or double valve replacement and coronary artery bypass grafting

Exclusion Criteria:

* Patients unable to give informed consent
* Patients younger than 18 years of age or older than 80 years
* Pregnancy or breastfeeding
* Ejection fraction (EF) of less than 30% preoperatively
* Preexisting renal insufficiency with a glomerular filtration rate below 30ml/min
* Patients transferred form the intensive care unit to the operating theater
* Emergency operation
* Reoperation
* Patients planned for fast-track surgery
* Patients planned for minimal extracorporal circuits
* Preexisting anemia requiring immediate perioperative blood transfusion
* Chronic inflammatory diseases
* Any signs of infection or sepsis
* Limitation of full therapy (e.g. Jehowa's witnesses)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2017-10-19 (Actual); Study Completion 2017-10-19 (Actual)

PRIMARY OUTCOMES:
Cumulative dose of inopressors (norepinephrine and epinephrine) per kg bodyweight/hour during the perioperative period | Perioperative period (induction of anesthesia until extubation in the intensive care unit, usually less than 24 hours))

SECONDARY OUTCOMES:
Time on inopressors | Perioperative period (induction of anesthesia until extubation in the intensive care unit, usually less than 24 hours))
Cumulative dose of inodilators | Perioperative period (induction of anesthesia until extubation in the intensive care unit, usually less than 24 hours))
Time on inodilators | Perioperative period (induction of anesthesia until extubation in the intensive care unit, usually less than 24 hours))
Cumulative dose of vasodilatators | Perioperative period (induction of anesthesia until extubation in the intensive care unit, usually less than 24 hours))
Time on vasodilatators | Perioperative period (induction of anesthesia until extubation in the intensive care unit, usually less than 24 hours))
Total amount of fluid | Perioperative period (induction of anesthesia until extubation in the intensive care unit, usually less than 24 hours))
Changes in acid-base status | Perioperative period (induction of anesthesia until extubation in the intensive care unit, usually less than 24 hours))

CONTACTS AND LOCATIONS:
Overall Officials: Carmen A Pfortmueller, MD, Principal Investigator — Department of Intensive Care, Bern University Hospital and University of Bern, Bern, Switzerland
Locations (1):
- Department of Intensive Care, Bern University Hospital and University of Bern, Bern, Switzerland, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pfortmueller CA, Faeh L, Muller M, Eberle B, Jenni H, Zante B, Prazak J, Englberger L, Takala J, Jakob SM. Fluid management in patients undergoing cardiac surgery: effects of an acetate- versus lactate-buffered balanced infusion solution on hemodynamic stability (HEMACETAT). Crit Care. 2019 May 6;23(1):159. doi: 10.1186/s13054-019-2423-8. PMID 31060591